CLINICAL TRIAL: NCT00922532
Title: Inhaled Nitric Oxide For The Treatment Of Hypoxic Respiratory Failure With Pulmonary Hypertension In Preterm Infants
Brief Title: Inhaled Nitric Oxide (INO) In Hypoxic Respiratory Failure
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision not to pursue prior to submission
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IK-3001-HRF-301
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Hypoxic Respiratory Failure With Pulmonary Hypertension
Keywords: Hypoxic Respiratory Failure (HRF), Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Inhaled Nitric Oxide (Experimental): Inhaled Nitric Oxide
  Interventions: Drug: Inhaled Nitric Oxide
- Nitrogen (Placebo Comparator): Nitrogen Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Inhaled Nitric Oxide will be administered continuously starting at 20ppm through an INOvent delivery system for up to 14 days.
  Other Names: INOmax
  Arms: Inhaled Nitric Oxide
Drug: Placebo — Nitrogen gas will be administered in the same manor as the experimental drug
  Arms: Nitrogen

SUMMARY:
This Phase 3, Double-blind, Randomized, Placebo controlled, multicenter study is to confirm the efficacy of inhaled nitric oxide for the management of hypoxic respiratory failure associated with pulmonary hypertension in preterm infants.

Study subjects will be administered either inhaled nitric oxide or placebo to determine if there is a change in oxygenation.

DETAILED DESCRIPTION:
This trial will be a multi-center, double blind, placebo-controlled, randomized clinical trial. All mothers identified with prolonged rupture of membranes and/or oligohydramnios, and all inborn infants < 30 weeks gestational age (GA) at birth will be screened for enrollment. Infants who meet all inclusion and exclusion criteria within the first 48 hours after birth will be randomized to either inhaled NO starting at 20 ppm, or matched placebo, delivered by means of a blinded INOvent® delivery device. Randomization will be stratified by center and treatment will be assigned using an interactive voice or web-based response system (IVRS). All infants will receive up to 14 days of therapy, following a dose reduction schedule. The primary outcome measure will be change in oxygenation at 1 hour after start of therapy. In order to determine the effects of iNO therapy on survival and need for mechanical ventilation, cross-over will not be allowed.

This clinical trial will attempt to demonstrate if pre-term infants may benefit from treatment with nitric oxide for inhalation. A multi-center study is necessary to recruit an appropriate number of subjects, and to reflect the variability of standard practice across the different participating centers. All treatment assignments are blinded in order to minimize the risk of bias in treatment and data collection. In addition, a concurrent placebo group has been chosen as the most appropriate control group since there may be temporal, institutional and national variations in average outcomes. Methemoglobin levels will be measured locally and will collected in a blinded manner.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants who:

* Are in-born at < 30 weeks gestational age
* Weigh 500-1250 grams
* Have hypoxic respiratory failure requiring mechanical ventilation with FiO2 > 0.8 to maintain SaO2 ≥ 85% in the first 48 hours after birth after use of exogenous surfactant
* Have minimal parenchymal lung disease by chest X ray

Exclusion Criteria:

Preterm infants who:

* Have ten minute Apgar score < 5
* Have life-threatening anomalies (cardiac, thoracic, chromosomal) or congenital diaphragmatic hernia with lung hypoplasia, or any child who will not receive complete intensive care
* Have bilateral Grade IV Intraventricular Hemorrhage (IVH)
* Are dependent on right to left shunting to maintain the systemic circulation
* Have received prior iNO therapy
* Have had treatment with investigational medications

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Arterial Blood Gases | Day 1 through Day 6

SECONDARY OUTCOMES:
Methemoglobin levels | Treatment Duration
Vital Signs | Study Duration
Adverse Events | Study Duration
cGMP Levels | Day 1 through 14